CLINICAL TRIAL: NCT00919399
Title: Phase II Study Evaluating the Effectiveness of the Exemestane (Aromasin) With Tamoxifen on the Rate of Clinical Response Menopausal in Patients With Locally Advanced Breast Tumors
Brief Title: Exemestane (Aromasine) + Tamoxifen - Breast Neo-Adjuvant
Acronym: TAMARO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: PHARMACIA SAS (Unknown)
Responsible Party: Henri Roché - Professor, Institut Claudius Regaud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01 SEIN 03
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; locally advanced; Menopausal patient; aromasin; tamoxifen; efficacy
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Exemestane — 25mg a day during 4 months
  Other Names: AROMASINE®
Drug: tamoxifen — One 20 mg tablet a day started 1 week after the first Aromasine intake
  Other Names: KESSAR®

SUMMARY:
This is a Phase II non-randomized, open, uncontrolled and bi-centric study of hormonal induction by exemestane (Aromasin) + tamoxifen to evaluate the effectiveness of exemestane (Aromasin) with tamoxifen on the rate of clinical response menopausal in patients with tumors of locally advanced breast. Hormone therapy will be administered at a dose of 25mg/day for exemestane and 20 mg / day for 4 months for tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer histologically proven by a 14 G or 16 G micro-biopsy to have confirmation of the diagnosis, evaluation histology prognosis grade, hormone receptors and to obtain a sample for the study of biological factors.
* Menopausal patients as defined as follows:

  * Natural menopause >= 1 year, or
  * Surgical ovariectomy.
* T unilateral tumor> 3 cm, N 1-2, M0 or M +, non-inflammatory.
* Hormone receptor positive. RE positive or PR positive with histochemical technique (+ 10% of cells express the receptor)
* No previous treatment of the disease by chemotherapy, hormone therapy, surgery or radiotherapy. Discontinuation of replacement therapy of menopause for at least 1 month
* Age>= 60 years
* Evaluable disease
* Performance Status <= 2
* Biological function using the following criteria:

  * neutrophils >= 2.10E9 / l,
  * Platelets> = 100.10E9 / l,
  * Hemoglobin> = 10 g / dl,
  * Creatinine <= 1.5 x upper normal,
  * Total bilirubin <= 1.25 x the upper normal
  * Transaminases (AST and ALT) <= 1.5 x upper normal,
  * Alkaline phosphatase <= 2.5 x upper normal.
* Cardiac Function: electrocardiogram (ECG) normal.
* Signed written consent before any procedure related to the study.

Exclusion Criteria:

* Men
* Non Menopausal Patients
* Patients with hormone receptor negative: PR- and RE -
* Contra-indication to anti-estrogens (risk thrombi arteria)
* Tumor <3 cm operable
* Tumor inflammatory T4d (PEV 2 or 3).
* Extensive hepatic lesions (> 1 / 3 of liver volume)
* Uncontrolled cardiac disease such as angina, congestive heart failure, or arrhythmia requiring medical treatment or history of myocardial infarction within 3 months before.
* History of cancer except skin cancer and basal cell cancer in situ of the cervix (a contralateral breast cancer had been no systemic treatment will be admitted).
* Chronic diseases (somatic or psychiatric) in poor prognosis.
* Patients who for reasons of family, social, geographical or psychological can not be followed properly.
* Patients under law protection

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the objective response rate (complete response and partial response) | June 2006

SECONDARY OUTCOMES:
Pharmacokinetic interaction between Exemestane and Tamoxifen | june 2006

CONTACTS AND LOCATIONS:
Overall Officials: Henri ROCHE, Principal Investigator — Institut Claudius Regaud
Locations (2):
- France (2):
  - CHU de Toulouse Rangueil, Toulouse
  - Institut Claudius Regaud, Toulouse